CLINICAL TRIAL: NCT06626165
Title: Mirikizumab Therapy is Effective for Patients With Moderate to Severe Ulcerative Colitis Patients Whose Geboes Score Grade is ≥3.2) on Endoscopic Biopsy
Brief Title: Association Between Effectiveness of Mirikizumab and UC Patients With High Neutrophilic Infiltration in Epithelium of the Colonic Mucosa
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Showa Inan General Hospital (Other)
Responsible Party: Principal Investigator, Akira Horiuchi, Chief, Digestive Disease Center, Showa Inan General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Geboes 3.2
Record Dates: First submitted 2024-07-20; First posted 2024-10-03 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2024-09

CONDITIONS: Ulcerative Colitis
Keywords: ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — mirikizumab; vedolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Mirikizumab (Active Comparator): When the patients were endoscopically active and pathologically high neutrophil infiltration in epithelium of the colonic mucosa (Geboes score Grade ≥3.2), using Geboes biopsy histology scores they will be administered by mirikizumab.
  Interventions: Drug: Mirikizumab
- Vedolizumab (Active Comparator): When the patients are endoscopically active and pathologically low neutrophil infiltration in epithelium of the colonic mucosa (Geboes score Grade 3.1), using Geboes biopsy histology scores, they will be administered by vedolizumab.
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Mirikizumab — Mirikizmgab will be administered based on the result of Geboes score Grade ≥ 3.2.
  Arms: Mirikizumab
Drug: Vedolizumab — Vedolizmab will be administered based on the result of Geboes score Grade 3.1.
  Arms: Vedolizumab

SUMMARY:
The goal of this study is to confirm that Mirikizumab therapy may provide clinical, endoscopic, and histopathologic improvements in patients with moderate to severe UC refractory to maintenance therapy when high neutrophilic infiltration in epithelium of the colonic mucosa (Geboes score Grade ≥3.2) on endoscopic biopsy is found.

ELIGIBILITY:
Inclusion Criteria:

* They were endoscopically active ulcerative colitis patients.

Exclusion Criteria:

* the presence of a long-term illness, colorectal cancer, or infectious colitis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-07-20 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Changes in clinical activities before and after mirikizumab or vedolizumab treatment. | 2 weeks
  Clinical activity is graded using the clinical activity index (0, best - 15, worst).

SECONDARY OUTCOMES:
Changes in endoscopic activities before and after mirikizumab or vedolizumab administration. | 2 months
  Mayo endoscopic subscore (0, best - 3, worst) and ulcerative colitis endoscopic index of severity (UCEIS) score are assessed at the site with the maximum endoscopic activity, (0, best - 8, worst).
Changes in pathological activity | 2 months
  Pathological activity was graded using Geboes biopsy histology scores, which were classified on a scale from 0 to 5, with higher scores indicating more severe histologic inflammation.

CONTACTS AND LOCATIONS:
Locations (1):
- Showa Inan General Hospital, Komagane, Nagano, Japan

IPD SHARING:
Plan to Share IPD: Undecided